CLINICAL TRIAL: NCT06244849
Title: TOward a Better Understanding of the autoPhagy Machinery for the Identification of Potential Novel Biomarkers and Therapeutic Targets in Crohn's Disease - TOPIC Study
Acronym: TOPIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Centre International de Recherche en Infectiologie (CIRI) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL22_1172
Record Dates: First submitted 2023-12-14; First posted 2024-02-06 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Crohn's Disease
Keywords: Crohn disease; Autophagy flux; Intestinal microbiota; Biomarker; Non-inflammatory bowel diseases
MeSH Terms: conditions — Crohn Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: A case-control study from a prospective bicentric cohort of CD patients. Proof of concept and exploratory study with minimum risks (type 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with Crohn disease (n=150) (Other): CD patients requiring to undergo an ileo-colonoscopy for routine investigations (assessment of disease activity or complications as stricture or screening of colorectal cancer for CD)
  Interventions: Biological: Blood samples; Biological: Stool simple; Biological: Ileocolonic biopsies
- Patient without Crohn disease (n=20) (Other): Non-IBD patients (control) requiring to undergo an ileo-colonoscopy for routine investigations (screening for colorectal cancer or diagnosis of irritable bowel syndrome for controls).
  Interventions: Biological: Blood samples; Biological: Stool simple; Biological: Ileocolonic biopsies

INTERVENTIONS:
Biological: Blood samples — A 28 mL (5 EDTA tubes of 4 mL and 2 dry tubes) venous blood will be collected added to the standard blood analysis performed in routine
Biological: Stool simple — A fresh stool sample will be collected and conserved at room temperature until shipment
Biological: Ileocolonic biopsies — An ileo-colonoscopy with 10 ileal biopsies scheduled in their regular medical follow-up will be performed

SUMMARY:
Crohn's disease (CD) belongs to chronic inflammatory bowel diseases (IBD) affecting over 2 million individuals in the North America and 3.2 million in Europe with an increasing incidence rate in newly industrialized countries experiencing a westernization of lifestyle (1). This highly disabling disease affects patients' life in several ways with severe complications requiring surgery for half of them and is responsible for considerable economic burdens (2,3). Decades of research displayed that CD pathogenesis is determined by inappropriate immune responses towards luminal microbiota in genetically susceptible hosts. Genome-wide association studies (GWAS) have identified autophagy as one of the main pathways associated with susceptibility to CD (4-6). Autophagy is a dynamic process of the lysosomal catabolism, called autophagy flux, which is crucial to degrade and recycle obsolete and deleterious cytosolic components of the cell (7). Autophagy is also the main cell-autonomous process to fight intracellular microorganisms by degrading them, and by contributing to antimicrobial host immune responses. However, the functional consequences of polymorphisms affecting autophagy-associated genes on the dynamic process of autophagy and its real impact on CD pathogenesis remain largely unknown. In addition, CD is associated with a gut microbiota dysbiosis, as exemplified by the higher prevalence of AIEC (a bacterium eliminated by autophagy) in ileal mucosa of CD patients (8-10). Hence, autophagy defect, linked to autophagy SNPs, could contribute to CD-related dysbiosis and to CD activity and severity.

Beyond, CD-associated abnormalities of the autophagy flux may affect the composition of the autophagic cargoes, as well as the one of other vesicular pathway, such as exosomes, known to influence autophagy. These impairments could affect at longer term both cell activities and immune responses, especially in antigen presenting cells, which drive host immune responses.

The TOPIC project concerns translational research, in which we plan to generate a prospective cohort of CD patients giving up the unique opportunity to collect clinical data, to analyse simultaneously the autophagy flux, genetic variants of interest (from blood samples) and intestinal microbiota (from intestinal samples) and allowing to perform more fundamental studies. The results of the fundamental part will allow a better understanding of the pathophysiology of CD, and ultimately better management of these patients.

ELIGIBILITY:
--- Inclusion Criteria :

For CD patients :

* Aged over 18 years
* Men or non-pregnant women
* Patients with a diagnosis of terminal ileum or ileocolonic CD for at least three months who requires to perform an ileocolonoscopy for routine follow-up
* Inactive and moderately to severely active CD according to the Harvey-Bradshaw index
* Stable doses of oral prednisone (≤30 mg per day) or budesonide (≤9 mg per day), mesalamine, concomitant immunosuppressive agents, biologics including anti-TNF agents, vedolizumab or ustekinumab are allowed at stable dose for at least three months before inclusion.
* Informed written consent
* Beneficiary or beneficiary of a social security system

For non IBD controls :

* Aged over 18 years
* Men or non-pregnant women
* Patients without a diagnosis of Crohn's disease who requires to perform an ileocolonoscopy for routine follow-up
* Informed written consent
* Beneficiary or beneficiary of a social security system

  * Exclusion Criteria * :

For patients and non-IBD controls :

* Existing pregnancy, lactation, or intended pregnancy within the next 15 months
* History of disease, including mental/emotional disorder that might interfere with their participation in the study
* Serious secondary illnesses of an acute or chronic nature, which in the opinion of the investigator renders the patient unsuitable for inclusion into the study
* Inability to comply with the protocol requirements
* Presence of an ileo-/colonic stoma
* Patients with known colonic stricture and exclusive or predominant anal or perineal Crohn's disease lesions
* Known previous or concurrent malignancy (other than that considered surgically cured, with no evidence for recurrence for 5 years)
* Short bowel syndrome
* Concomitant Clostridium difficile superinfection
* Indeterminate colitis
* Concomitant leukocyte apheresis
* Patients who will be exposed to antibiotics 4 weeks prior the inclusion, given the potential impact on the detection of AIEC colonization in ileal biopsies
* Patients who denied the protocol, not ability to accept or sign consent of the protocol
* Subject involved in another interventional research with an exclusion period still in progress at inclusion
* Pregnant women, women in labor or breastfeeding women*.
* Persons deprived of their liberty by a judicial or administrative decision
* Persons under psychiatric care
* Persons admitted to a health or social institution for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Subject involved in another clinical trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Autophagy flux | Baseline and the day of ileocolonoscopy
  Difference of the autophagy flux signature according to AIEC infection, autophagy related gene variants, and its relationship between CD activity and severity.

SECONDARY OUTCOMES:
Characterize and compare the autophagosomal proteome in CD genetic autophagicvariant expressing immune cells in ileum and in colon in CD patients from that in non IBD patients (controls). | Baseline and the day of ileocolonoscopy
  Qualitative and/or quantitative comparative analysis of content of the autophagosomal cargos between CD patients expressing the CD-associated autophagy related variants and WT gene-expressing non-IBD controls.
Characterize and compare the exosomal proteome in CD genetic autophagic variant expressing immune cells in ileum and in colon in CD patients from that in non IBD patients (controls). | Baseline and the day of ileocolonoscopy
  Qualitative and/or quantitative comparative analysis of content of the exosomal proteome cargos between CD patients expressing the CD-associated autophagy related variants and WT gene-expressing non-IBD controls.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Estaing, Clermont-Ferrand
  - Centres Hospitalier Lyon Sud, Pierre-Bénite

IPD SHARING:
Plan to Share IPD: Undecided